CLINICAL TRIAL: NCT04999969
Title: A Phase II Study to Evaluate the Safety, Pharmacokinetics, and Clinical Activity of AZD0171 in Combination With Durvalumab and Chemotherapy in Participants With Locally Advanced or Metastatic Solid Tumours
Brief Title: Safety, Pharmacokinetics and Clinical Activity of AZD0171 in Combination With Durvalumab and Chemotherapy in Locally Advanced or Metastatic Solid Tumours
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D8151C00001; 2021-002040-78 (EudraCT Number)
Record Dates: First submitted 2021-08-03; First posted 2021-08-11 (Actual); Results first posted 2025-11-26 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced or Metastatic Solid Tumours
Keywords: AZD0171; Durvalumab; Gemcitabine; Nab-paclitaxel; Leukaemia inhibitory factor; Pancreatic ductal adenocarcinoma; Immunotherapy
MeSH Terms: interventions — durvalumab; Gemcitabine; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AZD0171 + Durvalumab + chemotherapy (Experimental): Participants will receive AZD0171 (intravenous [IV]) along with durvalumab (IV) in combination with standard-of-care chemotherapy IV (gemcitabine and nab-paclitaxel).
  Interventions: Drug: AZD0171; Drug: Durvalumab; Drug: Gemcitabine; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: AZD0171 — AZD0171
  Other Names: MSC-1
Drug: Durvalumab — Durvalumab
  Other Names: MEDI4736
Drug: Gemcitabine — Chemotherapy (Standard-of-Care)
Drug: Nab-paclitaxel — Chemotherapy (Standard-of-Care)

SUMMARY:
The proposed study is designed to examine the effects of AZD0171 and durvalumab in combination with standard-of-care chemotherapy in patients with pancreatic ductal adenocarcinoma (PDAC).

DETAILED DESCRIPTION:
This is a Phase II, open-label, single arm, multicentre study to assess the safety, preliminary antitumour activity, immunogenicity, pharmacodynamics (PD), and pharmacokinetics (PK) of AZD0171 in combination with durvalumab and standard-of-care chemotherapy (gemcitabine and nab-paclitaxel) in participants with first line (1L) metastatic pancreatic ductal adenocarcinoma (mPDAC).

All participants will be treated until progressive disease or unacceptable toxicity or withdrawal of consent or another discontinuation criterion is met.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group performance status of 0 or 1 at screening/enrolment
* Must have a Gustave Roussy Immune Score of 0 or 1
* Participants diagnosed with histologically confirmed metastatic pancreatic adenocarcinoma
* Participants must have at least 1 measurable lesion to be called a target lesion according to RECIST v1.1
* All participants must consent to providing sufficient archival specimen taken during metastatic stage or fresh tumour specimens for tumoural CD8+ T cell testing for enrolment
* Presence of tumoural CD8+ T cells based on a predetermined benchmarked PDAC external sample
* Normal organ and bone marrow function measured within 28 days prior to first dose of study intervention
* Body weight ≥ 35 kg

Exclusion Criteria:

* Symptomatic central nervous system metastasis or any history of leptomeningeal disease or cord compression
* A participant with an already known sensitising mutation or tumour characteristic for pancreatic cancer for which there is a preferred local standard-of-care treatment
* History of thromboembolic event within the past 3 months prior to the scheduled first dose of study intervention
* Any unresolved toxicities ≥ Grade 2 per Common Terminology Criteria for Adverse Events v5.0 from prior therapy (excluding vitiligo, alopecia, controlled diabetes)
* History of solid organ transplantation
* History of active primary immunodeficiency
* Ongoing or an active infection, including tuberculosis, hepatitis B, hepatitis C, or human immunodeficiency virus. A negative COVID-19 PCR test taken within 28 days of the start of the study treatment is required.
* Uncontrolled intercurrent illness
* Participants with prior history of myocardial infarction, transient ischemic attack, coronary bypass, or stroke within the past 3 months prior to the first dose of study intervention
* Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated from 3 electrocardiograms
* Active or prior documented autoimmune or inflammatory disorders
* History of another primary malignancy
* Receipt of any conventional or investigational anticancer therapy prior to the scheduled first dose of study intervention
* Prior receipt of any immune-mediated therapy
* Use of immunosuppressive medication within 14 days prior to the first dose of study intervention
* Receipt of live, attenuated vaccine within 28 days prior to the first dose of study intervention (Participants can receive non-live COVID-19 vaccines, at the discretion of the Investigator)

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2024-10-07 (Actual); Study Completion 2026-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (16):
  - Research Site, La Jolla, California
  - Research Site, Los Angeles, California
  - Research Site, Orange, California
  - Research Site, Ventura, California
  - Research Site, Atlanta, Georgia
  - Research Site, Coeur d'Alene, Idaho
  - Research Site, Boston, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Grand Rapids, Michigan
  - Research Site, Buffalo, New York
  - Research Site, New York, New York
  - Research Site, Portland, Oregon
  - Research Site, San Antonio, Texas
  - Research Site, Charlottesville, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Madison, Wisconsin
- Canada (2):
  - Research Site, Barrie, Ontario
  - Research Site, Toronto, Ontario
- South Korea (2):
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (5):
  - Research Site, Badalona
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Pamplona

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8151C00001&attachmentIdentifier=e7b04e49-2ac7-41d1-9909-8772adced022&fileName=258542_Redacted_CSP_Final_PDF.pdf&versionIdentifier=
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8151C00001&attachmentIdentifier=dfaea5fa-b524-4325-8b02-e6f497820249&fileName=258542_Redacted_CSR_Synopsis_Final_PDF.pdf&versionIdentifier=
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8151C00001&attachmentIdentifier=4f2e8e34-5b4c-4710-be00-39f3a52ff50d&fileName=258542_Redacted_SAP_Final_PDF.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled participants across 39 sites in 4 countries. The enrollment period began on December 10, 2021, and the analyses presented in this form are based on clinical data lock date of November 16, 2024.
Pre-assignment Details: Participants who met the inclusion criteria and none of the exclusion criteria were enrolled to the study. All the study assessments were performed as per the schedule of assessment.
Groups:
- AZD0171 + Durvalumab + Chemotherapy: Participants received AZD0171 (intravenous [IV]) along with durvalumab IV in combination with standard-of-care chemotherapy IV (gemcitabine and nab-paclitaxel) until disease progression, death, lost to follow-up or consent withdrawal which ever occurred first.
Period: Overall Study
Arm/Group | AZD0171 + Durvalumab + Chemotherapy
Started | 126
Completed | 41
Not Completed | 85
Not completed — Death | 76
Not completed — Progressive Disease | 1
Not completed — Withdrawal by Subject | 8

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) set, which included all participants who received any dose of study treatment.
Arm/Group | AZD0171 + Durvalumab + Chemotherapy
Number analyzed (Participants) | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 71
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 4
  Native Hawaiian or Other Pacific Islander | 0
  American Indian or Alaska Native | 0
  Asian | 21
  White | 94
  Other | 1
  Not Reported | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 110
  Unknown | 0
  Missing | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs), Immune Mediated AEs (imAEs) and Serious AEs (SAEs)
Description: The safety and tolerability of study intervention (AZD0171, durvalumab, and standard-of-care chemotherapy) was assessed. The grading scales found in the revised National Cancer Institute CTCAE latest version was utilized for all events with an assigned CTCAE grading. Grade refers to the severity of the AE. The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL. Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living (ADL); Grade 4: Life-threatening, urgent intervention required; Grade 5: Death related to AE.
Time Frame: From Cycle 1 Day 1 (each cycle was 28 days in length) until Day 90 (post last dose of study intervention), up to 34 months
Population: Safety set, which included all participants who received any amount of study treatment.
  As specified in the below data table, in the row entitled, 'Any AE leading to dose reduction of AZD0171', one participant had recorded one reduced dose event of AZD0171 by error. This event was not a dose reduction; but, the study treatment was interrupted due to an AE of infusion related reaction, therefore only partial dose was administered.
Measure: Count of Participants; unit: Participants
Arm/Group | AZD0171 + Durvalumab + Chemotherapy
Number analyzed (Participants) | 126
Participants
  Any AE | 126
  Any AE possibly related to treatment | 123
  Any AE possibly related to AZD0171 | 99
  Any AE possibly related to Durvalumab | 107
  Any AE possibly related to Nab-paclitaxel | 123
  Any AE possibly related to Gemcitabine | 122
  Any AE of >= Common Terminology Criteria for Adverse Events (CTCAE) grade 3 | 115
  Any AE of >= CTCAE grade 3, possibly related to treatment | 90
  Any AE of >= CTCAE grade 3, possibly related to AZD0171 | 46
  Any AE of >= CTCAE grade 3, possibly related to Durvalumab | 45
  Any AE of >= CTCAE grade 3, possibly related to Nab-paclitaxel | 82
  Any AE of >= CTCAE grade 3, possibly related to Gemcitabine | 84
  Any SAE (Serious Adverse Event) | 72
  Any SAE possibly related to treatment | 30
  Any SAE possibly related to AZD0171 | 14
  Any SAE possibly related to Durvalumab | 17
  Any SAE possibly related to Nab-paclitaxel | 20
  Any SAE possibly related to Gemcitabine | 21
  Any SAE of >= CTCAE grade 3 | 70
  Any SAE of >= CTCAE grade 3, possibly related to treatment | 27
  Any SAE of >= CTCAE grade 3, possibly related to AZD0171 | 11
  Any SAE of >= CTCAE grade 3, possibly related to Durvalumab | 16
  Any SAE of >= CTCAE grade 3, possibly related to Nab-paclitaxel | 16
  Any SAE of >= CTCAE grade 3, possibly related to Gemcitabine | 17
  Any SAE with outcome death | 15
  Any SAE with outcome death, possibly related to treatment | 3
  Any SAE with outcome death, possibly related to AZD0171 | 3
  Any SAE with outcome death, possibly related to Durvalumab | 2
  Any SAE with outcome death, possibly related to Nab-paclitaxel | 3
  Any SAE with outcome death, possibly related to Gemcitabine | 3
  Any AE leading to discontinuation of treatment | 37
  Any AE leading to discontinuation of AZD0171 | 32
  Any AE leading to discontinuation of Durvalumab | 31
  Any AE leading to discontinuation of Nab-paclitaxel | 31
  Any AE leading to discontinuation of Gemcitabine | 32
  Any AE leading to discontinuation of treatment, possibly related to treatment | 22
  Any AE leading to discontinuation of AZD0171, possibly related to AZD0171 | 11
  Any AE leading to discontinuation of Durvalumab, possibly related to Durvalumab | 12
  Any AE leading to discontinuation of Nab-paclitaxel, possibly related to Nab-paclitaxel | 9
  Any AE leading to discontinuation of Gemcitabine, possibly related to Gemcitabine | 11
  Any AE leading to drug interruption of treatment | 103
  Any AE leading to drug interruption of AZD0171 | 86
  Any AE leading to drug interruption of Durvalumab | 61
  Any AE leading to drug interruption of Nab-paclitaxel | 98
  Any AE leading to drug interruption of Gemcitabine | 94
  Any AE leading to dose reduction of treatment | 67
  Any AE leading to dose reduction of AZD0171 | 1
  Any AE leading to dose reduction of Durvalumab | 0
  Any AE leading to dose reduction of Nab-paclitaxel | 60
  Any AE leading to dose reduction of Gemcitabine | 54
  Any AE leading to dose modification of treatment | 110
  Any AE leading to dose modification of AZD0171 | 86
  Any AE leading to dose modification of Durvalumab | 61
  Any AE leading to dose modification of Nab-paclitaxel | 106
  Any AE leading to dose modification of Gemcitabine | 100
  Any SAE leading to discontinuation of treatment | 28
  Any SAE leading to discontinuation of AZD0171 | 27
  Any SAE leading to discontinuation of Durvalumab | 28
  Any SAE leading to discontinuation of Nab-paclitaxel | 26
  Any SAE leading to discontinuation of Gemcitabine | 27
  Any SAE leading to discontinuation of treatment, possibly related to treatment | 13
  Any SAE leading to discontinuation of AZD0171, possibly related to AZD0171 | 7
  Any SAE leading to discontinuation of Durvalumab, possibly related to Durvalumab | 10
  Any SAE leading to discontinuation of Nab-paclitaxel, possibly related to Nab-paclitaxel | 5
  Any SAE leading to discontinuation of Gemcitabine, possibly related to Gemcitabine | 6
  Any SAE leading to drug interruption of treatment | 36
  Any SAE leading to drug interruption of AZD0171 | 33
  Any SAE leading to drug interruption of Durvalumab | 24
  Any SAE leading to drug interruption of Nab-paclitaxel | 34
  Any SAE leading to drug interruption of Gemcitabine | 35
  Any SAE leading to dose reduction of treatment | 2
  Any SAE leading to dose reduction of AZD0171 | 0
  Any SAE leading to dose reduction of Durvalumab | 0
  Any SAE leading to dose reduction of Nab-paclitaxel | 2
  Any SAE leading to dose reduction of Gemcitabine | 2
  Any SAE leading to dose modification of treatment | 36
  Any SAE leading to dose modification of AZD0171 | 33
  Any SAE leading to dose modification of Durvalumab | 24
  Any SAE leading to dose modification of Nab-paclitaxel | 34
  Any SAE leading to dose modification of Gemcitabine | 35
  Any SAE leading to hospitalisation | 71
  Any immune mediated AEs | 45
  Any infusion reaction AEs | 11

2. Primary Outcome: Overall Survival at 12 Months (OS-12)
Description: Percentage of participants alive at 12 months after initiation of study intervention per Kaplan- Meier estimate of OS at 12 months.
Time Frame: At 12 months
Population: The ITT set, which included all participants who received any dose of study treatment.
Measure: Number (80% Confidence Interval); unit: Percentage
Arm/Group | AZD0171 + Durvalumab + Chemotherapy
Number analyzed (Participants) | 126
Percentage | 53.8 [47.79 to 59.50]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: The ORR is defined as the percentage of participants with a confirmed best overall response of complete response (CR) or partial response (PR) that occurred prior to the initiation of subsequent anti-cancer treatment and prior to progression. The ORR was assessed per Response Evaluation Criteria in Solid Tumours (RECIST) v1.1.
Time Frame: From Cycle 1 Day 1 (each cycle was 28 days in length) until initiation of subsequent anti-cancer treatment and prior to progression (up to 35 months).
Population: Response Evaluable Set (RES), which included all participants who had measurable disease at baseline.
Measure: Number (80% Confidence Interval); unit: Percentage
Arm/Group | AZD0171 + Durvalumab + Chemotherapy
Number analyzed (Participants) | 126
Percentage | 34.9 [29.30 to 40.91]

4. Secondary Outcome: Disease Control Rate (DCR)
Description: The DCR is defined as the percentage of participants with a best overall response of confirmed CR or PR, or who had stable disease (SD) maintained for 16 weeks from first dose. DCR was assessed per RECIST v1.1 criteria.
Time Frame: Up to 16 weeks
Population: The ITT set, which included all participants who received any dose of study treatment.
Measure: Number (80% Confidence Interval); unit: Percentage
Arm/Group | AZD0171 + Durvalumab + Chemotherapy
Number analyzed (Participants) | 126
Percentage | 65.9 [59.90 to 71.46]

5. Secondary Outcome: Duration of Response (DoR)
Description: The DoR is defined as the time from first documented objective response (confirmed CR or confirmed PR) until date of first documented disease progression or death (by any cause in the absence of disease progression). The DoR was assessed per RECIST v1.1 criteria.
Time Frame: From screening until disease progression or last evaluable assessment in the absence of progression, whichever came first (up to 35 months)
Population: The ITT set, which included all participants who received any dose of study treatment.
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | AZD0171 + Durvalumab + Chemotherapy
Number analyzed (Participants) | 126
Months | 7.72 [6.439 to 9.462]

6. Secondary Outcome: Median Progression Free Survival (PFS)
Description: The PFS is defined as the time from first dose of study intervention until the date of objective disease progression or death (by any cause in the absence of progression), whichever was earlier. The PFS was analyzed using the Kaplan-Meier method.
Time Frame: From first dose of study intervention until disease progression or last evaluable assessment in the absence of progression, whichever came first (up to 35 months)
Population: The ITT set, which included all participants who received any dose of study treatment.
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | AZD0171 + Durvalumab + Chemotherapy
Number analyzed (Participants) | 126
Months | 7.33 [6.801 to 7.918]

7. Secondary Outcome: Progression Free Survival at 4 Months (PFS-4)
Description: The percentage of participants alive and free of progression at 4 months per Kaplan-Meier estimate.
Time Frame: At 4 months
Population: The ITT set, which included all participants who received any dose of study treatment.
Measure: Number (80% Confidence Interval); unit: Percentage
Arm/Group | AZD0171 + Durvalumab + Chemotherapy
Number analyzed (Participants) | 126
Percentage | 75.5 [69.95 to 80.13]

8. Secondary Outcome: Median Overall Survival (OS)
Description: The OS is defined as the time from the start of study intervention to the date of death due to any cause.
Time Frame: From first dose of study intervention until death (Up to 35 months) or from first dose of study intervention until last evaluable assessment (Up to 35 months)
Population: The ITT set, which included all participants who received any dose of study treatment.
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | AZD0171 + Durvalumab + Chemotherapy
Number analyzed (Participants) | 126
Months | 13.67 [11.565 to 15.639]

9. Secondary Outcome: Change From Baseline in Serum Levels of Carbohydrate Antigen 19-9 (CA19-9)
Description: Mean change from baseline was assessed for serum CA19-9
Time Frame: Day 1 of each Cycle through Cycle 27 (each cycle was 28 days in length), at end of treatment and at Day 28 follow up (post last dose); up to 35 months
Population: The Pharmacodynamic (PD) set, which included all participants who received any amount of study treatment with at least one reportable PD measurement. The number analyzed "n" refers to the number of participants included in analysis in specific time points.
Measure: Mean (Standard Deviation); unit: Units/milliliter (U/mL)
Arm/Group | AZD0171 + Durvalumab + Chemotherapy
Number analyzed (Participants) | 126
Units/milliliter (U/mL)
  Cycle 01 Day 01: number analyzed (Participants) | 6
  Cycle 01 Day 01 | 0.0 (0.0)
  Cycle 02 Day 01: number analyzed (Participants) | 109
  Cycle 02 Day 01 | -12717.2 (95596.8)
  Cycle 03 Day 01: number analyzed (Participants) | 103
  Cycle 03 Day 01 | -17463.4 (99400.5)
  Cycle 04 Day 01: number analyzed (Participants) | 91
  Cycle 04 Day 01 | -19283.0 (106081.2)
  Cycle 05 Day 01: number analyzed (Participants) | 86
  Cycle 05 Day 01 | -19823.2 (109490.0)
  Cycle 06 Day 01: number analyzed (Participants) | 77
  Cycle 06 Day 01 | -21974.6 (115724.1)
  Cycle 07 Day 01: number analyzed (Participants) | 66
  Cycle 07 Day 01 | -25249.6 (124848.3)
  Cycle 08 Day 01: number analyzed (Participants) | 61
  Cycle 08 Day 01 | -26902.4 (129722.0)
  Cycle 09 Day 01: number analyzed (Participants) | 46
  Cycle 09 Day 01 | -12230.2 (31705.4)
  Cycle 10 Day 01: number analyzed (Participants) | 39
  Cycle 10 Day 01 | -570.9 (29271.1)
  Cycle 11 Day 01: number analyzed (Participants) | 30
  Cycle 11 Day 01 | -3363.4 (6647.6)
  Cycle 12 Day 01: number analyzed (Participants) | 28
  Cycle 12 Day 01 | -3469.5 (6766.1)
  Cycle 13 Day 01: number analyzed (Participants) | 19
  Cycle 13 Day 01 | -2674.8 (6895.7)
  Cycle 14 Day 01: number analyzed (Participants) | 18
  Cycle 14 Day 01 | -3100.1 (6768.7)
  Cycle 15 Day 01: number analyzed (Participants) | 13
  Cycle 15 Day 01 | -1229.7 (2027.1)
  Cycle 16 Day 01: number analyzed (Participants) | 7
  Cycle 16 Day 01 | -1346.8 (2040.8)
  Cycle 17 Day 01: number analyzed (Participants) | 6
  Cycle 17 Day 01 | -1470.2 (2171.6)
  Cycle 18 Day 01: number analyzed (Participants) | 4
  Cycle 18 Day 01 | -1867.5 (2666.0)
  Cycle 19 Day 01: number analyzed (Participants) | 4
  Cycle 19 Day 01 | -1868.8 (2691.3)
  Cycle 20 Day 01: number analyzed (Participants) | 3
  Cycle 20 Day 01 | -1928.7 (3255.2)
  Cycle 21 Day 01: number analyzed (Participants) | 4
  Cycle 21 Day 01 | -1830.8 (2663.2)
  Cycle 22 Day 01: number analyzed (Participants) | 3
  Cycle 22 Day 01 | -1903.7 (3244.6)
  Cycle 23 Day 01: number analyzed (Participants) | 3
  Cycle 23 Day 01 | -1854.3 (3240.4)
  Cycle 24 Day 01: number analyzed (Participants) | 2
  Cycle 24 Day 01 | -2764.5 (3909.6)
  Cycle 25 Day 01: number analyzed (Participants) | 1
  Cycle 25 Day 01 | 0.9 (NA) — Standard deviation is not calculable due to insufficient number of participants
  Cycle 26 Day 01: number analyzed (Participants) | 1
  Cycle 26 Day 01 | 0 (NA) — Standard deviation is not calculable due to insufficient number of participants
  Cycle 27 Day 01: number analyzed (Participants) | 1
  Cycle 27 Day 01 | 0 (NA) — Standard deviation is not calculable due to insufficient number of participants
  End of treatment: number analyzed (Participants) | 79
  End of treatment | -471.3 (145796.2)
  Day 28 Follow up: number analyzed (Participants) | 52
  Day 28 Follow up | 19574.2 (114348.1)

10. Secondary Outcome: Number of Participants With Positive Anti-drug Antibodies (ADAs) Against AZD0171 in Serum
Description: Number and percentage of participants in the below categories are provided:(i)ADA positive (+ve) at baseline and/or post-baseline visits. The percentage of these participants in a population is known as ADA prevalence(ii)ADA +ve post-baseline and not detected at baseline (treatment-induced ADA positive)(iii)Treatment-boosted ADA +ve:Baseline +ve ADA titre-boosted to a 4-fold or higher level following drug administration(iv)Treatment-emergent ADA +ve:The sum of treatment-induced ADA +ve and treatment-boosted ADA +ve. The percentage of these participants in a population is known as ADA incidence(v)Persistent +ve:ADA negative (-ve) at baseline and having at least 2 post-baseline ADA +ve measurements with ≥ 16 weeks between first and last positive, or an ADA +ve result at the last available post-baseline assessment(vi)Transient +ve:ADA -ve at baseline and at least 1 post-baseline ADA +ve measurement and not fulfilling the conditions for persistently +ve.
Time Frame: Cycle 1 (Days 1 and 15), Cycle 2 (Days 1 and 15), until Day 90 post last dose of study intervention (each cycle is 28 days in length), assessed up to 35 months
Population: Immunogenicity set, which included all participants who received at least one dose of investigational product (IP) with at least one reportable immunogenicity assessment. The number analyzed "n" refers to the number of participants included in analysis of specific ADA category as mentioned below, [a] Participants with ADA result at baseline and/or post-baseline [b] Participants with ADA result at baseline and ≥1 post-baseline [c] Participants with ADA result at baseline only.
Measure: Count of Participants; unit: Participants
Arm/Group | AZD0171 + Durvalumab + Chemotherapy
Number analyzed (Participants) | 126
Participants
  ADA positive at baseline and/or post-baseline (ADA prevalence) (a) | 2
  Treatment Emergent-ADA positive AZD0171: number analyzed (Participants) | 116
  Treatment Emergent-ADA positive AZD0171 | 0
  Treatment-induced ADA positive (b): number analyzed (Participants) | 116
  Treatment-induced ADA positive (b) | 0
  Treatment-boosted ADA positive (b): number analyzed (Participants) | 116
  Treatment-boosted ADA positive (b) | 0
  Both baseline and post-baseline positive (b): number analyzed (Participants) | 116
  Both baseline and post-baseline positive (b) | 0
  Only baseline positive (c): number analyzed (Participants) | 116
  Only baseline positive (c) | 0
  ADA persistently positive (b): number analyzed (Participants) | 116
  ADA persistently positive (b) | 0
  ADA transiently positive (b): number analyzed (Participants) | 116
  ADA transiently positive (b) | 0

11. Secondary Outcome: Number of Participants With Positive Anti-drug Antibodies (ADAs) Against Durvalumab in Serum
Description: as for outcome 10
Time Frame: as for outcome 10
Population: Immunogenicity set, which included all participants who received at least one dose of IP with at least one reportable immunogenicity assessment. The number analyzed "n" refers to the number of participants included in analysis of specific ADA category as mentioned below, [a] Number of participants with ADA result at baseline and/or post-baseline [b] Number of participants with ADA result at baseline and ≥1 post-baseline [c] Number of participants with ADA result at baseline only.
Measure: Count of Participants; unit: Participants
Arm/Group | AZD0171 + Durvalumab + Chemotherapy
Number analyzed (Participants) | 126
Participants
  ADA positive at baseline and/or post-baseline (ADA prevalence) (a) | 8
  Treatment Emergent-ADA positive (ADA incidence) (b): number analyzed (Participants) | 116
  Treatment Emergent-ADA positive (ADA incidence) (b) | 0
  Treatment-induced ADA positive (b): number analyzed (Participants) | 116
  Treatment-induced ADA positive (b) | 0
  Treatment-boosted ADA positive (b): number analyzed (Participants) | 116
  Treatment-boosted ADA positive (b) | 0
  Both baseline and post-baseline positive (b): number analyzed (Participants) | 116
  Both baseline and post-baseline positive (b) | 0
  Only baseline positive (c): number analyzed (Participants) | 116
  Only baseline positive (c) | 3
  ADA persistently positive (b): number analyzed (Participants) | 116
  ADA persistently positive (b) | 0
  ADA transiently positive (b): number analyzed (Participants) | 116
  ADA transiently positive (b) | 0

12. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of AZD0171
Description: The maximum concentration of AZD0171 was determined.
Time Frame: Cycle 1 Day 1 and Cycle 4 Day 1 (each cycle is 28 days in length)
Population: The PK set which included all participants who received any amount of study treatment with at least one reportable PK measurement. The number analyzed, 'n', refers to participants with intensive PK sampling at specific time points, who were included in the noncompartmental analysis (NCA). Additional population PK/PK analyses are available under reference: 39041713.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/mililiter (ug/mL)
Arm/Group | AZD0171 + Durvalumab + Chemotherapy
Number analyzed (Participants) | 9
microgram/mililiter (ug/mL)
  Cycle 01 Day 01 | 395.4 (16.84)
  Cycle 04 Day 01: number analyzed (Participants) | 3
  Cycle 04 Day 01 | 694.6 (31.62)

13. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Nab-paclitaxel
Description: The Cmax of Nab-paclitaxel was determined.
Time Frame: Cycle 1 Day 15 and Cycle 4 Day 15 (each cycle is 28 days in length)
Population: The PK set which included all participants who received any amount of study treatment with at least one reportable PK measurement. The number analyzed, 'n', refers to participants with intensive PK sampling at specific time points, who were included in the NCA. Additional population PK/PK analyses are available under reference: 39041713.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/mililiter (ng/ml)
Arm/Group | AZD0171 + Durvalumab + Chemotherapy
Number analyzed (Participants) | 6
nanogram/mililiter (ng/ml)
  Cycle 01 Day 15 | 1996 (176.4)
  Cycle 04 Day 15: number analyzed (Participants) | 4
  Cycle 04 Day 15 | 1113 (553.2)

14. Secondary Outcome: Area Under Plasma Concentration-time Curve From Zero to Infinity (AUCinf) of AZD0171
Description: The AUCinf of AZD0171 was determined.
Time Frame: Cycle 1 Day 1 (each cycle is 28 days in length)
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | AZD0171 + Durvalumab + Chemotherapy
Number analyzed (Participants) | 9
h*ug/mL | 56570 (77.33)

15. Secondary Outcome: Area Under the Concentration-time Curve From Zero to the Last Quantifiable Concentration (AUClast) of AZD0171
Description: The AUClast of AZD0171 was determined.
Time Frame: Cycle 1 Day 1 and Cycle 4 Day 1 (each cycle is 28 days in length)
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | AZD0171 + Durvalumab + Chemotherapy
Number analyzed (Participants) | 9
h*ug/mL
  AUClast Cycle 01 Day 01 | 38600 (87.50)
  AUClast Cycle 04 Day 01: number analyzed (Participants) | 3
  AUClast Cycle 04 Day 01 | 66290 (44.47)

16. Secondary Outcome: Area Under the Concentration-time Curve From Zero to the Last Quantifiable Concentration (AUClast) of Nab-paclitaxel
Description: The AUClast of Nab-paclitaxel was determined.
Time Frame: Cycle 1 Day 15 and Cycle 4 Day 15 (each cycle is 28 days in length)
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram/milliliter (h*ng/mL)
Arm/Group | AZD0171 + Durvalumab + Chemotherapy
Number analyzed (Participants) | 6
hour*nanogram/milliliter (h*ng/mL)
  AUClast Cycle 01 Day 15 | 3992 (63.70)
  AUClast Cycle 04 Day 15: number analyzed (Participants) | 4
  AUClast Cycle 04 Day 15 | 2853 (107.7)

17. Secondary Outcome: Area Under the Concentration-time Curve in the Dose Interval (AUCtau) of AZD0171
Description: The AUCtau of AZD0171 was determined.
Time Frame: Cycle 1 Day 1 and Cycle 4 Day 1 (each cycle is 28 days in length)
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*microgram/milliliter (h*ug/mL)
Arm/Group | AZD0171 + Durvalumab + Chemotherapy
Number analyzed (Participants) | 9
hour*microgram/milliliter (h*ug/mL)
  AUCtau Cycle 01 Day 01 | 43770 (55.76)
  AUCtau Cycle 04 Day 01: number analyzed (Participants) | 2
  AUCtau Cycle 04 Day 01 | 81760 (14.11)

18. Secondary Outcome: Area Under the Concentration-time Curve in the Dose Interval (AUCtau) of Nab-paclitaxel
Description: The AUCtau of Nab-paclitaxel was determined.
Time Frame: Cycle 1 Day 15 and Cycle 4 Day 15 (each cycle is 28 days in length)
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram/milliliter (h*ng/mL)
Arm/Group | AZD0171 + Durvalumab + Chemotherapy
Number analyzed (Participants) | 6
hour*nanogram/milliliter (h*ng/mL)
  AUCtau Cycle 01 Day 15 | 4550 (54.03)
  AUCtau Cycle 04 Day 15: number analyzed (Participants) | 4
  AUCtau Cycle 04 Day 15 | 3302 (98.07)

19. Secondary Outcome: Clearance (CL) of AZD0171
Description: The CL of AZD0171 was determined.
Time Frame: Cycle 1 Day 1 and Cycle 4 and Day 1 (each cycle is 28 days in length)
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/hour (L/h)
Arm/Group | AZD0171 + Durvalumab + Chemotherapy
Number analyzed (Participants) | 9
Liter/hour (L/h)
  Cycle 01 Day 01 | 0.02651 (77.33)
  Cycle 04 Day 01: number analyzed (Participants) | 2
  Cycle 04 Day 01 | 0.01835 (14.11)

20. Secondary Outcome: Clearance (CL) of Nab-paclitaxel
Description: The CL of Nab-paclitaxel was determined.
Time Frame: Cycle 1 Day 15 and Cycle 4 Day 15 (each cycle is 28 days in length)
Population: PK set which included all participants who received any amount of study treatment with at least one reportable PK measurement. The number analyzed, 'n', refers to participants with intensive PK sampling at specific time points, who were included in the NCA. Additional population PK/PK analyses are available under reference: 39041713.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/hour/meter square (L/h/m**2)
Arm/Group | AZD0171 + Durvalumab + Chemotherapy
Number analyzed (Participants) | 6
Liter/hour/meter square (L/h/m**2)
  Cycle 1 Day 15 | 51.37 (67.48)
  Cycle 4 Day 15: number analyzed (Participants) | 4
  Cycle 4 Day 15 | 67.13 (99.70)

21. Secondary Outcome: Terminal Elimination Half-life (t1/2λz) of AZD0171
Description: The t1/2λz of AZD0171 was determined.
Time Frame: Cycle 1 Day 1 and Cycle 4 Day 1 (each cycle is 28 days in length)
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | AZD0171 + Durvalumab + Chemotherapy
Number analyzed (Participants) | 9
Hours
  Cycle 01 Day 01 | 127.4 (77.48)
  Cycle 04 Day 01: number analyzed (Participants) | 2
  Cycle 04 Day 01 | 188.2 (6.567)

22. Secondary Outcome: Terminal Elimination Half-life (t1/2λz) of Nab-paclitaxel
Description: The t1/2λz of Nab-paclitaxel was determined.
Time Frame: Cycle 1 Day 15 and Cycle 4 Day 15 (each cycle is 28 days in length)
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | AZD0171 + Durvalumab + Chemotherapy
Number analyzed (Participants) | 6
Hours
  Cycle 1 Day 15 | 7.353 (85.14)
  Cycle 4 Day 15: number analyzed (Participants) | 4
  Cycle 4 Day 15 | 9.509 (20.20)

23. Secondary Outcome: Change From Screening in Cluster of Differentiation 8 (CD8+) T Cell Tumour Infiltration in Central Tumour Region
Description: The changes in CD8+ T cell tumour infiltration (on-treatment during cycle 3 minus baseline) associated with AZD0171 treatment in combination with durvalumab and chemotherapy was assessed in participants with 1L metastatic pancreatic ductal adenocarcinoma.
Time Frame: In cycle 3 (each cycle was 28 days in length), subsequent to the first disease assessment scan conducted at roughly 8 weeks.
Population: The PD set, which included all participants who received any amount of study treatment with at least one reportable PD measurement. The number analyzed "n" refers to the number of participants included in analysis in specific time points.
Measure: Mean (Standard Deviation); unit: Cells/millimeter square
Arm/Group | AZD0171 + Durvalumab + Chemotherapy
Number analyzed (Participants) | 23
Cells/millimeter square
  Central tumor region | 2.86 (378.12)
  Central tumor region - within Pan-cytokeratin (PanCK)- Tumor Stroma Area | -10.66 (460.92)
  Central tumor region- within PanCK+ Carcinoma Cell Compartment | -25.68 (329.00)

24. Secondary Outcome: Serum Concentration of Total Leukaemia Inhibitory Factor (LIF) Over Time
Description: Serum concentration of LIF bound to AZD0171 (total LIF) was assessed.
Time Frame: Cycle 1 Day 1 and Day 15, Cycle 2 Day 1 and Day 15, Cycle 3 Day 1 and Day 15, Cycle 4 Day 1 and Day 15, Cycle 5Day 1, Cycle 6 Day 1, Cycle 7 Day 1, Cycle 8 Day 1 and Cycle 11 Day 1 (each cycle is 28 days in length)
Population: The PD set, which included all participants who received any amount of study treatment with at least one reportable PD measurement. The number analyzed, 'n', refers to participants with intensive PK sampling at specific time points, who were included in the NCA. Additional population PK/PK analyses are available under reference: 39041713.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram/millilitre (pg/mL)
Arm/Group | AZD0171 + Durvalumab + Chemotherapy
Number analyzed (Participants) | 126
picogram/millilitre (pg/mL)
  Cycle 01 Day 01: number analyzed (Participants) | 5
  Cycle 01 Day 01 | 82.01 (55.91)
  Cycle 01 Day 15: number analyzed (Participants) | 19
  Cycle 01 Day 15 | 284.6 (93.92)
  Cycle 02 Day 01: number analyzed (Participants) | 32
  Cycle 02 Day 01 | 195.5 (85.89)
  Cycle 02 Day 15: number analyzed (Participants) | 28
  Cycle 02 Day 15 | 174.9 (69.12)
  Cycle 03 Day 01: number analyzed (Participants) | 26
  Cycle 03 Day 01 | 201.4 (106.4)
  Cycle 03 Day 15: number analyzed (Participants) | 21
  Cycle 03 Day 15 | 169.2 (63.66)
  Cycle 04 Day 01: number analyzed (Participants) | 23
  Cycle 04 Day 01 | 166.2 (59.66)
  Cycle 04 Day 15: number analyzed (Participants) | 25
  Cycle 04 Day 15 | 139.5 (71.98)
  Cycle 05 Day 01: number analyzed (Participants) | 25
  Cycle 05 Day 01 | 169.2 (71.97)
  Cycle 06 Day 01: number analyzed (Participants) | 5
  Cycle 06 Day 01 | 182.5 (96.65)
  Cycle 07 Day 01: number analyzed (Participants) | 1
  Cycle 07 Day 01 | 310.0 (NA) — Standard deviation is not calculable due to insufficient number of participants
  Cycle 08 Day 01: number analyzed (Participants) | 14
  Cycle 08 Day 01 | 187.8 (94.74)
  Cycle 11 Day 01: number analyzed (Participants) | 6
  Cycle 11 Day 01 | 133.2 (50.24)

ADVERSE EVENTS:
Time Frame: From Cycle 1 Day 1 (each cycle was 28 days in length) until Day 90 (post last dose of study intervention), up to 34 months.
Description: All adverse events during the trial are reported.
Arm/Group | AZD0171 + Durvalumab + Chemotherapy
All-Cause Mortality (participants affected / at risk) | 76/126
Serious Adverse Events (participants affected / at risk) | 72/126
Other Adverse Events (participants affected / at risk) | 126/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD0171 + Durvalumab + Chemotherapy (N=126)
Colitis (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Duodenal obstruction (Gastrointestinal disorders) | 4 (7)
Gastritis erosive (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2)
Intestinal perforation (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 2 (2)
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 3 (4)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 3 (4)
Asthenia (General disorders) | 2 (2)
Chills (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pyrexia (General disorders) | 4 (5)
Sudden death (General disorders) | 1 (1)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1)
Biliary obstruction (Hepatobiliary disorders) | 2 (2)
Cholangitis (Hepatobiliary disorders) | 5 (6)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Cholangitis acute (Hepatobiliary disorders) | 1 (2)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 3 (3)
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 2 (2)
Appendicitis perforated (Infections and infestations) | 1 (1)
Bacteraemia (Infections and infestations) | 3 (3)
Biliary tract infection (Infections and infestations) | 4 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Covid-19 (Infections and infestations) | 1 (1)
Catheter site infection (Infections and infestations) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Haemophilus infection (Infections and infestations) | 1 (1)
Hepatic infection (Infections and infestations) | 3 (3)
Liver abscess (Infections and infestations) | 1 (1)
Necrotising fasciitis (Infections and infestations) | 1 (1)
Pancreatic abscess (Infections and infestations) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 6 (6)
Pneumonia aspiration (Infections and infestations) | 1 (2)
Sepsis (Infections and infestations) | 14 (15)
Septic shock (Infections and infestations) | 2 (2)
Urosepsis (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 3 (3)
Toxic encephalopathy (Nervous system disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Hypertensive urgency (Vascular disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Shock (Vascular disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD0171 + Durvalumab + Chemotherapy (N=126)
COVID-19 (Infections and infestations) | 13 (13)
Candida infection (Infections and infestations) | 7 (7)
Urinary tract infection (Infections and infestations) | 12 (21)
Anaemia (Blood and lymphatic system disorders) | 62 (99)
Leukocytosis (Blood and lymphatic system disorders) | 7 (7)
Neutropenia (Blood and lymphatic system disorders) | 27 (59)
Thrombocytopenia (Blood and lymphatic system disorders) | 21 (37)
Hypothyroidism (Endocrine disorders) | 7 (7)
Decreased appetite (Metabolism and nutrition disorders) | 43 (60)
Dehydration (Metabolism and nutrition disorders) | 15 (21)
Hyperglycaemia (Metabolism and nutrition disorders) | 13 (14)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 10 (11)
Hypokalaemia (Metabolism and nutrition disorders) | 17 (25)
Hypomagnesaemia (Metabolism and nutrition disorders) | 13 (21)
Hyponatraemia (Metabolism and nutrition disorders) | 11 (12)
Insomnia (Psychiatric disorders) | 15 (17)
Dizziness (Nervous system disorders) | 23 (29)
Dysgeusia (Nervous system disorders) | 34 (36)
Headache (Nervous system disorders) | 18 (20)
Neuropathy peripheral (Nervous system disorders) | 24 (25)
Neurotoxicity (Nervous system disorders) | 9 (13)
Peripheral motor neuropathy (Nervous system disorders) | 7 (7)
Peripheral sensory neuropathy (Nervous system disorders) | 41 (44)
Sinus tachycardia (Cardiac disorders) | 7 (8)
Deep vein thrombosis (Vascular disorders) | 8 (8)
Hypertension (Vascular disorders) | 15 (19)
Hypotension (Vascular disorders) | 16 (17)
Cough (Respiratory, thoracic and mediastinal disorders) | 16 (17)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 23 (31)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 13 (15)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Abdominal distension (Gastrointestinal disorders) | 7 (7)
Abdominal pain (Gastrointestinal disorders) | 41 (52)
Abdominal pain upper (Gastrointestinal disorders) | 7 (8)
Constipation (Gastrointestinal disorders) | 31 (39)
Diarrhoea (Gastrointestinal disorders) | 73 (126)
Dry mouth (Gastrointestinal disorders) | 10 (12)
Dyspepsia (Gastrointestinal disorders) | 9 (10)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 8 (9)
Nausea (Gastrointestinal disorders) | 69 (110)
Stomatitis (Gastrointestinal disorders) | 16 (23)
Vomiting (Gastrointestinal disorders) | 41 (77)
Alopecia (Skin and subcutaneous tissue disorders) | 45 (48)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 17 (18)
Erythema (Skin and subcutaneous tissue disorders) | 8 (9)
Pruritus (Skin and subcutaneous tissue disorders) | 26 (29)
Rash (Skin and subcutaneous tissue disorders) | 12 (16)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 26 (34)
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 (17)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 15 (17)
Myalgia (Musculoskeletal and connective tissue disorders) | 16 (21)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 (18)
Asthenia (General disorders) | 37 (77)
Chills (General disorders) | 12 (17)
Fatigue (General disorders) | 63 (90)
Influenza like illness (General disorders) | 10 (11)
Mucosal inflammation (General disorders) | 11 (11)
Oedema peripheral (General disorders) | 48 (75)
Pyrexia (General disorders) | 55 (126)
Alanine aminotransferase increased (Investigations) | 38 (54)
Aspartate aminotransferase increased (Investigations) | 32 (51)
Blood alkaline phosphatase increased (Investigations) | 7 (8)
Gamma-glutamyltransferase increased (Investigations) | 12 (12)
Neutrophil count decreased (Investigations) | 42 (80)
Platelet count decreased (Investigations) | 19 (33)
Weight decreased (Investigations) | 20 (24)
White blood cell count decreased (Investigations) | 13 (19)
Fall (Injury, poisoning and procedural complications) | 8 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No unpublished information may be disclosed without prior written approval from AstraZeneca.

DOCUMENTS (2):
  • Study Protocol (2024-05-03): https://cdn.clinicaltrials.gov/large-docs/69/NCT04999969/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-26): https://cdn.clinicaltrials.gov/large-docs/69/NCT04999969/SAP_001.pdf